CLINICAL TRIAL: NCT00562237
Title: Randomized, Observer-Blind, Placebo-Controlled Study to Assess the Immunogenicity and Safety of Two Adjuvant Formulations of an Egg-Derived Pandemic Surface Antigen Influenza Vaccine in Healthy Adults Aged ≥18 Years and ≤ 49 Years.
Brief Title: Immunogenicity and Safety of Two Adjuvant Formulations of an Egg-Derived Pandemic Vaccine
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This trial discontinued on 20 JUN 2008 because the interim immunogenicity results do not justify these formulations as pandemic vaccine candidates
Sponsor: Solvay Pharmaceuticals (Industry)
Responsible Party: Joost Melis, Solvay Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: S205.1.001; 2007-000876-17
Record Dates: First submitted 2007-11-20; First posted 2007-11-21 (Estimated); Last update posted 2008-10-27 (Estimated); Status verified 2008-10

CONDITIONS: Healthy Subjects
Keywords: immunogenicity; safety; adjuvanted pandemic vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- 1 (Placebo Comparator)
  Interventions: Biological: S205 placebo
- 2 (Experimental)
  Interventions: Biological: S205 10ugHA
- 3 (Experimental)
  Interventions: Biological: S205 30ugHA
- 4 (Experimental)
  Interventions: Biological: S205 10ugHA+500ugAlOH
- 5 (Experimental)
  Interventions: Biological: S205 30ugHA+500ugAlOH
- 6 (Experimental)
  Interventions: Biological: S205 10ugHA+1250ugAlOH
- 7 (Experimental)
  Interventions: Biological: S205 30ugHA+1250ugAlOH

INTERVENTIONS:
Biological: S205 placebo — 2 i.m. injections per subject (0.5 mL each)
  Arms: 1
Biological: S205 10ugHA — 2 i.m. injections per subject (0.5 mL each)
  Arms: 2
Biological: S205 30ugHA — 2 i.m. injections per subject (0.5 mL each)
  Arms: 3
Biological: S205 10ugHA+500ugAlOH — 2 i.m. injections per subject (0.5 mL each)
  Arms: 4
Biological: S205 30ugHA+500ugAlOH — 2 i.m. injections per subject (0.5 mL each)
  Arms: 5
Biological: S205 10ugHA+1250ugAlOH — 2 i.m. injections per subject (0.5 mL each)
  Arms: 6
Biological: S205 30ugHA+1250ugAlOH — 2 i.m. injections per subject (0.5 mL each)
  Arms: 7

SUMMARY:
Several combinations of H5N1 antigen concentrations and aluminium-hydroxide adjuvant concentrations will be tested for their safety and capacity to induce a specific immune response.

ELIGIBILITY:
Inclusion Criteria:

* being healthy and ≥ 18 and ≤ 49 years of age
* willing and able to give informed consent

Exclusion Criteria:

* having participated in an influenza H5 vaccine trial in the past
* known to be allergic to any constituent of the vaccine
* serious adverse reactions to previous (influenza) vaccination
* currently participating in another clinical trial or having participated in any clinical trial in the month preceding the start of the study
* using medication that influences the immune system

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2007-07; Primary Completion 2007-11 (Actual); Study Completion 2008-09 (Estimated)

PRIMARY OUTCOMES:
Hemagglutination inhibition titers | one year

SECONDARY OUTCOMES:
CHMP criteria | one year
Virus neutralization | one year
Anti-HA antibody level kinetics | one year
Safety | one year

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (6):
- Finland (3):
  - Site 21, Helsinki
  - Site 22, Tampere
  - Site 23, Turku
- Germany (3):
  - Site 12, Goch
  - Site 10, Hamburg
  - Site 11, Nuremberg